CLINICAL TRIAL: NCT01363518
Title: Operative Versus Nonoperative Treatment of Humeral Shaft Fractures: A Prospective Cohort Comparison Study
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: Boston Medical Center (Other); Inova Fairfax Hospital (Other); Indiana University (Other); Prisma Health-Midlands (Other); Vanderbilt University (Other); Wake Forest University (Other); University of North Carolina (Other); Lahey Clinic (Other)
Responsible Party: Principal Investigator, Howard Place, MD, Professor, St. Louis University
Other Study IDs: 16589
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Closed Fracture of Shaft of Humerus
Keywords: humerus; fracture; operative treatment; non-operative treatment
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Operative: Operative group would have had surgery to treat their broken humerus.
- Nonoperative: Nonoperative group would have been treated with a brace, no surgery.

SUMMARY:
The subject's broken humerus (arm) is suitable for treatment with a fracture brace or operative fixation with plate and screws. Both of these types of treatments are often used by doctors to fix broken bones. If the subject agrees to participate in this study, the subject will be assigned by the treating surgeon to one of the following groups:

Group B: Non-operative treatment with a fracture brace Group P: a plate & screws - a metal device placed on top of the bone.

The investigators will collect information about the subject's arm fracture as it is treated with examinations and X-rays. X-rays will be obtained often in the first several months, depending on how the fracture is healing. This is determined by the doctor and will not be determined by the subject's participation in this research study.

Both treatments are routinely used and this study hopes to provide information regarding each type of treatment on the subject's functional outcome. A subject's treatment will not be affected whether they choose to participate in this research study or not.

The treatment of these subjects is no different because of this study. The treating surgeon will discuss with the patient their preferred treatment for the isolated humeral shaft fracture. If they meet the inclusion/exclusion criteria, they will be approached for participation in one of two treatment groups depending on a previous decision by the patient and the treating surgeon.

Hypotheses:

1. Patients with an isolated humeral shaft fracture that are plated will have a more rapid return to ADL's, work and full functional capacity than patients treated conservatively.
2. Patients treated with plate technique will have a more rapid improvement in functional outcome scores, decreased pain scores and patient satisfaction than those managed conservatively.
3. Complication rates of infection and iatrogenic neurologic injury will be higher in patients treated operatively.
4. Nonunion and malunion will be higher in patients managed conservatively.

DETAILED DESCRIPTION:
A. Rationale Humeral shaft fractures (OTA 12A, B or C) are not uncommon injuries and have been long considered fractures, which respond well to conservative (or nonoperative) management. Since Bohler's (1964) statement that humeral shaft fractures are "the most benign of all fractures of the long bones", many additional peer-reviewed publications have concluded that conservative management of this injury, in isolation, produces an excellent and uncomplicated result. Sarmiento's work resulted in a treatment algorithm utilizing functional bracing which remains the accepted standard of care for isolated humeral shaft fractures. Much of the early work on operative treatment of this injury reflected results, often poor, obtained when utilizing early generation implants and surgical techniques. In addition, a number of studies have reported the results of humeral shaft fractures managed with intramedullary nails. Although controversy remains, we believe the publications of McCormack, et.al.1 and Chapman, et.al.2 have concluded in a prospective randomized comparison fashion that plating now produces a superior outcome to intramedullary nailing in humeral shaft fractures. Very few existing publications3-7 compare conservative versus operative treatment of humeral shaft fractures. Of these, only one (Nast-Kolb, et.al.3) does so in a prospective manner. Even this study included patients with various associated and possibly confounding injuries and treatment selection was not controlled or randomized in any way.

No study has ever compared the results of isolated humeral shaft fractures treated conservatively/nonoperatively versus operatively in a prospective cohort comparison. In addition, few studies of humeral shaft fractures have utilized any form of validated functional outcome measures when drawing conclusions about given treatment options.

B. Hypothesis or Objective The objective of this study is to determine whether isolated humeral shaft fractures are optimally treated with internal fixation or bracing.

Specific Aim #1 To determine the healing rates between operative and non operative management in a prospective study.

Hypothesis 1. Nonunion and malunion will be higher in patients managed conservatively.

Specific Aim #2 The DASH outcomes of patients treated operatively will return to pre-injury status faster than non operative treatment.

Hypothesis 2.Patients with an isolated humeral shaft fracture that is operatively stabilized will have improved functional outcome scores as measure by the DASH score than patients treated conservatively.

Specific Aim #3 To determine VAS derived pain scores. Hypothesis 3. Patients treated with operative fixation will have decreased pain scores as measure by a VAS at 2 and 6 weeks than those managed conservatively.

Specific Aim #4 To determine overall complication rates between the two groups. Hypothesis 4. Complication rates of infection and iatrogenic neurologic injury will be higher in patients treated operatively.

C. Research Strategy We believe the need for this study is further supported by published data obtained in a retrospective review of two hundred thirteen (213) closed humeral shaft fractures treated operatively with plates and nonoperatively at the two Level I trauma centers over the past five years. These findings indicate a higher malunion and nonunion rate of statistical significance in the nonoperative group.

We are completing a pilot prospective, randomized cohort study with 62 patients enrolled and 31 in each group. We believe a large, prospective randomized study to answer the question of the better treatment in terms of functional outcomes for the treatment of humeral shaft fractures is needed.

This investigation will consist of a prospective, surgeon based multicenter clinical trial to evaluate non-operative versus operative treatment of isolated humeral shaft fractures.

C1.Study Participants This investigation will consist of a prospective multicenter clinical trial to evaluate non-operative versus operative treatment of isolated humeral shaft fractures. We anticipate participation from multiple Level I trauma centers; each of which has experience with similar research study designs. The PI and Co-investigators all participated in the pilot study, along with investigators from 5 additional centers. The study protocol will require IRB/HAC approval from each participating center.

Patient Recruitment and Screening When a patient from 18-65 years old presents with a humeral shaft fracture, he or she will be screened for possible enrollment in the study using the inclusion/exclusion criteria. If the patient is deemed appropriate by the treating surgeon, meaning that they meet all the inclusion criteria and do not meet any exclusion criteria, the patient will be given the consent form to read and it will be reviewed with the patient with time allowed to answer all questions. If the patient agrees to enter the study, he or she will sign the consent form.

Randomization The patients who provide informed consent will be randomized to one of two treatment groups: Patients in the brace group (B) will be treated with a fracture brace and patients randomized to the plate group (P) will be treated with open reduction and internal fixation (ORIF) with a plate. Each arm of the study will be separately randomized via a computer-generated number at the Data Control Center.

Assessment. The DASH (Disabilities of the Arm, Shoulder and Hand) Outcome Measure will be utilized as the functional assessment tool. As this tool has been well validated for upper extremity injuries and has normative data, we believe it to be a good choice for this study population. The questionnaire will be administered (we will compare operative to non operative treatment, not to patient's baseline function) at 6 weeks, 3, 6 and 12 months post-injury. In addition a visual analogue pain scale (VAS) will be administered at 2 weeks, 6 weeks, 3, 6 and 12 months.

C2. Treatment Patient who present with a humeral shaft fracture will initially have the same treatment. All patients will have a closed reduction with adequate sedation in the Emergency Department and application of a coaptation splint and sling. If they meet the inclusion/exclusion criteria, they will be approached for participation in one of two treatment groups. Informed consent will be obtained.

Patients in the operative group (P) will be scheduled for elective surgery for plate fixation of their humeral shaft fracture within 2 weeks from date of injury. The surgical approach, plate brand, and plate size will be at the discretion of the treating orthopaedic surgeon.

Patients in the non-operative group (B) will have clinical follow-up scheduled. A humeral fracture brace is applied in the office. A sling is optional for patient comfort. After fracture brace application, the patient is instructed to perform pendulum exercises for shoulder mobility. Exercises of the elbow, wrist and hand are also encouraged. The patient is instructed to adjust the tension of the brace twice per week and sleep in a semi-erect position for the first six weeks. (These instructions are all standard of care for fracture brace treatment). The fracture brace is worn until the patient has met the clinical and radiographic healing criteria described in the protocol.

D. Research Area Although accepted standards for non-operative management of isolated humeral shaft fractures have remained largely unchanged and unchallenged for several decades; prospective, comparative data incorporating validated patient outcome measures is lacking. Specifically, data comparing non-operative versus operative treatment for isolated humeral shaft fractures has not been published. We endeavor to scientifically evaluate two different treatments for isolated humeral shaft fractures and determine which treatment option in a prospective study may provide better functional outcomes and less complications.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a closed, humeral shaft fracture
2. English Speaking
3. Age between 18-65 at the time of injury
4. Entry into the study within 2 weeks of injury
5. Available for follow-up for at least 12 months
6. Patient signs informed consent

Exclusion Criteria:

1. Age less than 18 or greater than 65 at time of injury
2. Patients who are skeletally immature
3. Humeral shaft fractures that extend into the articular surface
4. Open humeral shaft fractures
5. Additional long bone injuries of upper or lower extremity that would compromise outcome assessment
6. Vascular injury requiring repair
7. Pathologic fracture
8. Definitive treatment delay of more than 2 weeks from initial injury
9. Immunocompromised patient
10. Unable to comply with post-operative rehabilitation protocols or instructions
11. Current or impending incarceration
12. Unlikely to follow-up in surgeon's estimation
13. Pregnant or lactating female
14. Previous retained hardware in humeral shaft

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 years with a humeral shaft fracture.
Sampling Method: Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2010-05; Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is the Disability of Arm, Shoulder and Hand (DASH) score. | Enrollment, 12 Week, 6 Month, and 12 Month Follow-Ups
  10 units difference of DASH will be considered as a clinically meaning full difference. Based on previous studies, the standard deviation of DASH is around 20. With 64 subjects in each group (total 128), we will have 80% power to detect a difference in mean of 10 between two study arms assuming the common standard deviation is 20 using a student t-test with type I error rate 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Cannada, M.D., Principal Investigator — St. Louis University
Locations (7):
- United States (7):
  - Indiana University-Wishard Hospital, Indianapolis, Indiana
  - Boston University Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Fairfax, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No
Results will be shared